CLINICAL TRIAL: NCT06364020
Title: Assessment of Risk Factors in Patients With Non-carious Cervical Lesions
Acronym: LACIS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230067
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Anxiety; Stress; Non-carious Cervical Lesions
Keywords: Periodontics; Anxiety,; Gingival recession; Feeding and Eating disorders; Bruxism; Restorative dentistry; NonCarious Cervical Lesions
MeSH Terms: conditions — Anxiety Disorders; Gingival Recession; Feeding and Eating Disorders; Bruxism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients seen in specialized periodontology consultation at Rothschild Hospital: The population that will be studied will be patients received in the first specialized clinical periodontology consultation aged between 18 and 60 years.

SUMMARY:
In the management of patients with noncarious cervical lesions (NCCL), we observe that they frequently present signs of anxiety, traumatic brushing, bruxism or eating disorders. These multifactorial and interrelated etiologies make diagnosis and management difficult. Furthermore, in the literature, there is a lack of studies that evaluate the relationship between these risk factors and NCCL. A better understanding of the etiology and risk factors would help to optimize patient management and direct patients to the most appropriate therapies.

DETAILED DESCRIPTION:
Tooth wear is a cumulative loss of surface area at the expense of mineralized tooth tissue caused by physical or physicochemical processes (erosion, attrition, abrasion), i.e., excluding carious lesion, resorption, or trauma.

Non-carious cervical lesions (NCCL) correspond to hard tissue loss in the cervical area of the tooth by processes not related to caries.

The prevalence of NCCL varies between 5 and 85% depending on the study and the severity of cervical wear increases with age. A 2020 systematic review estimates the prevalence of NCCL at 46.7%.

NCCL are frequent pathologies caused by changes in lifestyle and diet. The reasons for consultation are diverse and varied, either symptomatic (sensitivities) functional (food retention) or aesthetic. The prevalence and severity of wear increases with age. It is generally accepted that lesions are not generated by a single factor but result from a combination of factors, such as erosion, abrasion or abfraction. The clinical appearance of NCCLs may vary depending on the type and severity of the etiologic factors involved. Proper diagnosis of this type of lesion requires a comprehensive knowledge of the different etiologies as well as their multifactorial aspects through focused questioning and careful clinical observation. Due to the multifactorial and interrelated etiologies, accurate diagnosis of NCCLs is challenging.

Prevention and proper management of NCCL requires an understanding of the etiology and risk factors related to mental disorders such as depression, stress and anxiety or pathological behaviors such as traumatic brushing or bruxism. Wear lesions can be aggravated by gastroesophageal reflux and eating disorders resulting from mental disorders that are devastating to dental tissue. The decision to monitor NCCLs rather than intervene should be based on the progression of the lesions and how they compromise the vitality, function, and aesthetics of the teeth.

During the management of patients with NCCL, we observe that they show signs of anxiety. Therefore, the objective is to assess the level of anxiety in patients with NCCL and to compare it to that of patients without NCCL.

We wish to carry out an observational survey from a prospective cohort at the Rothschild Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 60 years old;
* Specialized periodontal consultation.

Exclusion Criteria:

* Patients with co-morbidities that do not allow for adequate brushing of the teeth (Parkinson, Alzheimer...);
* Patients with removable prothesis for two years or more;
* Patients under guardianship or trusteeship.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients seen in specialized periodontology consultation at Rothschild Hospital.
  During the initial consultation, according to current protocol and practice, the practitioner performs a complete examination of the mouth and teeth and indicates in the patient's medical record the possible presence of oral pathologies, including the diagnosis of NCCL.
  The presence of NCCL is judged on all teeth and defined by the presence of 4 or more NCCLs with a depth (buccolingual) and height (occlusogingival) greater than or equal to 2 mm.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
To investigate the association between anxiety/stress and the presence of NCCL. | During inclusion visit
  Assessment questionnaire DASS21 (Depression Anxiety Stress (DASS-21 ; Lovibond & Lovibond, 1995).

SECONDARY OUTCOMES:
To investigate the association between bruxism and the presence of NCCL. | During inclusion visit
  SCOFF Questionnaire (Kutz et al. 2020)
To investigate the association between eating disorders and the presence of NCCL. | During inclusion visit
  Bruxism questionnaire (Khoury & al. 2016)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Mocquot, MCU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Rothschild - Service Odontologie, Paris, France

IPD SHARING:
Plan to Share IPD: No